CLINICAL TRIAL: NCT05799443
Title: Efficacy and Safety of SBRT Followed by Tislelizumab Plus Cetuximab and Irinotecan in Patients With Previously Treated RAS Wild-type Advanced Refractory Colorectal Cancer: a Phase II, Single-arm Study
Brief Title: Efficacy and Safety of SBRT Followed by Tislelizumab Plus Cetuximab and Irinotecan in Patients With Previously Treated RAS Wild-type Advanced Refractory Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEC
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT followed by tislelizumab plus cetuximab and irinotecan (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Irinotecan Hydrochloride; Drug: cetuximab; Radiation: SBRT

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab will be administered on day 1 of each cycle at 200mg once every 14 days.
Drug: Irinotecan Hydrochloride — Irinotecan will be administered on day 1 of each cycle at 180 mg/m2 once every 14 days.
Drug: cetuximab — cetuximab will be administered on day 1 of each cycle at 500 mg/m2 once every 14 days.
Radiation: SBRT — 8-10Gy×5F，QOD

SUMMARY:
To evaluate the efficacy and safety of SBRT followed by tislelizumab plus cetuximab and irinotecan in patients with previously treated RAS wild-type advanced refractory colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Physical Condition Score (ECOG PS) of the Eastern Cancer Cooperative Group (USA) 0 or 1;
* Colorectal cancer diagnosed histologically and/or cytologically has metastases or relapses that are not curable by surgery
* Have received first - and second-line systemic antitumor therapy for mCRC (chemotherapy drugs may include fluorouracil, oxaliplatin, irinotecan, e.g. XELOX, FOLFOX, FOLFIRI, FOLFOXIRI, XELIRI; Can be combined with or without targeted drugs, such as cetuximab, bevacizumab);And disease progression after second-line treatment;
* Evaluation of lung or liver metastases can be evaluated, with stereotactic radiotherapy maneuverability;
* At least one measurable lesion as defined in RECIST version 1.1;
* Fertile patients must be willing to take effective pregnancy avoidance measures during the study period and ≥120 days after the last dose; Female patients with negative urine or serum pregnancy test results within 7 days or less before the first administration of the study drug;
* Have fully understood this study and voluntarily signed informed consent.
* Adequate organ and bone marrow function, meeting the following definitions:

  1. Blood routine (no blood transfusion, no granulocyte colony stimulating factor [G-CSF], no other drug correction within 14 days before treatment);Absolute count of neutrophils (ANC) ≥1.5×109/L;Hemoglobin (HB) ≥9.0 g/dL;Platelet count (PLT) ≥80×109/L;
  2. Blood biochemistry, serum creatinine (Cr) ≤ 1.5× upper limit of normal (ULN) or creatinine clearance ≥60 mL/min;Serum albumin ≥2.8g/dL, for patients with poor nutritional status before neoadjuvant therapy, patients who met the requirements through parenteral nutrition could also be included in the group;Total bilirubin (TBIL) ≤ 1.5×ULN;Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤2.5×ULN;

Exclusion Criteria:

* 1. Pregnant or lactating women;
* Patients with a known history of allergy to any investigative drug, similar drug or excipient;
* Patients with risk of massive gastrointestinal bleeding or gastrointestinal obstruction;
* Patients with a history of thromboembolism, except thrombosis caused by PICC;
* There are patients with active infection;
* Patients with unmanageable hypertension (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90mmHg);
* Patients with brain metastases with clinical symptoms or imaging evidence;
* Contraindications exist in treatment with other chronic diseases;
* Patients with a history of immunotherapy-related myocarditis, pneumonia, colitis, hepatitis, nephritis, etc., with current AE ≥ grade 2;
* According to the evaluation criteria of NCI CTCAE version 5.0, there are patients with all kinds of toxicities ≥ grade 2 due to previous treatment;
* Other conditions that the researchers determined were not suitable for inclusion in the study.
* Received any antitumor therapy and participated in other clinical studies within 4 weeks before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-04-05 (Estimated); Primary Completion 2024-04-05 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From enrollment to 12 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | From enrollment to 12 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first
Overall Survival (OS) | From enrollment to 12 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death.

IPD SHARING:
Plan to Share IPD: No